CLINICAL TRIAL: NCT01605968
Title: A Comparative Efficacy and Safety Study Between BCT Silver Bandage and Aquacel® Ag. Dressing In Obstetrical and Gynecological Post-Op Wound Healing
Brief Title: A Comparative Efficacy and Safety Study Between Two Silver Containing Dressings In Post-Op Wound Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The rate of subject recruitment is too slow.
Sponsor: Bio-medical Carbon Technology Co., Ltd. (Industry)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS11176
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Surgical Wound
Keywords: Obstetrics; Gynecology; Wound healing
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCT Silver Bandage (Experimental)
  Interventions: Device: BCT Silver Bandage
- Aquacel® Ag. Dressing (Active Comparator)
  Interventions: Device: Aquacel® Ag. Dressing

INTERVENTIONS:
Device: BCT Silver Bandage — Activated carbon fiber impregnated with silver particles
  Arms: BCT Silver Bandage
Device: Aquacel® Ag. Dressing — Antimicrobial primary dressing incorporating the unique gelling action of Hydrofiber® Technology with ionic silver for wounds that are infected or at risk of infection.
  Arms: Aquacel® Ag. Dressing

SUMMARY:
Study objective:

The objective of this study is to evaluate through clinical criteria the clinical efficacy and safety of BCT Silver Bandage role in obstetrical and gynecological wound healing is as effective and safe as Aquacel® Ag. Dressing.

Study devices:

* Study device: BCT Silver Bandage
* Comparator device:"ConvaTec"Aquacel® Ag Hydrofiber Dressing

Study design:

* Randomized, Open-label, interventional, comparative, preventive study with Blinded evaluator.
* All subjects must meet all the inclusion & exclusion criteria to enter this study in pre-operative phase.
* Eligible subjects will be enrolled after a scheduled operative procedure.
* There is SEVEN visits in this study (one screening eligibility phase up to 7 days before OP day, and four post-op treatment scheduled visits consisting on 1st , 3rd day, 5th day, 12th day and two follow up visit on the 28th and the 42nd post-operative day.
* During each scheduled visit, each subject will have colored picture of his wound after dressing been removed, and on visit V6 for wound evaluation by blinded PI.

Number of subjects: It is expected to recruit ≧150 eligible subjects.

Study Duration: About eighteen month.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female of any race aged between 18 - 70 years old
* The subject is willing and able to understand, sign and date the study Informed Consent, and be able to adhere to the scheduled visits regimen.
* The subject is having surgery (Cesarean pfannenstiel or Open Laparotomy incision) within 1 week

Exclusion Criteria:

* Patients with known allergy or topical hypersensitivity to ionic silver or alginate
* Any systemic or local active dermatological disease that might interfere with the evaluation of the surgical site such as eczema, psoriasis, skin cancer, scleroderma, chronic urticarial
* Patients undergoing MRI (Magnetic Resonance Imaging) examination.
* Subject residence is outside the study center city
* Patients was participating in another clinical trial less than 30 days before participation in this trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Efficacy measurements | 42 days after operation
  1. Wound infection rate within 5 days after operation
  2. Wound healing evaluation by Stony Brook Scar Evaluation Scale (SBSES), to be evaluated by blinded PI at V6
  3. Skin discoloration around the incision wound and/or wound keloid formation rate at V6
  4. Patient and Observer Scar Assessment Scale (POSAS) on V3, V5 and V6

SECONDARY OUTCOMES:
Safety Measurement | 42 days after operation
  The incidence of postoperative skin reactions (defined as blisters, itching, erythematous change around the surgical wound site) within 5 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Jen Tseng, MD, Principal Investigator — Dep. of Gynecology and Obstetrics, Chung-Shan Medical University Hospital
Locations (1):
- Dep. of Gynecology and Obstetrics, Chung-Shan Medical University Hospital, Taichung, Taiwan